CLINICAL TRIAL: NCT01947101
Title: A Phase I Study of Fecal Microbiota Transplantation (FMT) in Immunomodulator Dependent Pediatric Ulcerative Colitis (UC)
Brief Title: Fecal Microbiota Transplantation (FMT) for Treatment of Ulcerative Colitis in Children
Acronym: FMT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Richard Kellermayer, Assistant Professor, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-30591; FMT- Ulcerative Colitis (Other: Internal)
Record Dates: First submitted 2013-09-13; First posted 2013-09-20 (Estimated); Last update posted 2016-06-14 (Estimated); Status verified 2016-06

CONDITIONS: Ulcerative Colitis
Keywords: Stool transplant; Ulcerative Colitis; Fecal transplant; Inflammatory Bowel Disease
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ulcerative Colitis (Experimental): Fecal Microbiota Transplant
  Interventions: Biological: Fecal Microbiota Transplant

INTERVENTIONS:
Biological: Fecal Microbiota Transplant — Fecal Microbiota Transplant will be endoscopically administered directly into the colon. Consecutive treatments will be given by rectal enema route.
  Other Names: stool transplant

SUMMARY:
Patients diagnosed with ulcerative colitis (UC), a specific type of inflammatory bowel disease, will be invited to take part in this study. The investigators do not know what causes UC. However, the microbes (such as bacteria and viruses), which normally live in our intestines are thought to play an important role in the development of UC. There are many treatment options for UC such as steroids,and other medications that decrease inflammation. However, none of these can cure the disease.

This study aims to treat pediatric UC in an alternative fashion by changing the microbes in the gut by giving the participant's stool specimens from healthy adult individuals. There is some evidence from a few cases of adult UC that this therapy may cure the disease or at least provide long lasting suppression (remission) of the symptoms. The investigators would like to test this therapeutic intervention in children with UC.

The purpose of this study is to (1) examine the microbiome of stool and colon (2) and to determine whether healthy-donated stool enemas can treat pediatric ulcerative colitis. (3) The investigators will also study the effects of the treatment on colonic gene expression.

DETAILED DESCRIPTION:
FMT RECIPIENTS:

Participants will be recruited from the patient population treated by the Pediatric Gastroenterology, Hepatology, and Nutrition Section at Baylor College of Medicine/Texas Children's Hospital.

I. Activities prior to starting FMT therapy:

1. Participants will be asked to discontinue or taper their current home medications for ulcerative colitis.
2. Participants will be asked to complete enema training.
3. The participant and family will be counseled in case emergency surgical and/or intensive care interventions are required.
4. Survey Completion to assess clinical symptoms.

II. Initiation of FMT Therapy:

1. Pre-colonoscopy and FMT therapy preparation:

   One to two days prior to scheduled colonoscopy the study participant will be asked to provide a stool sample. They will also undergo a bowel clean-out with Miralax for colonoscopy preparation. Colonoscopy (endoscopic examination of the large bowel) will be used to deliver the first donor fecal transplant at the beginning of the therapeutic protocol.
2. FMT treatment and Initial colonoscopy:

Fecal microbiota transplantation is made possible by utilizing a donor (healthy adult) providing their stool sample. The donor's stool will be screened and tested for known disease-causing agents including viruses, bacteria and parasites to prevent spread of disease to the participant.

On the first day of treatment, the participant will undergo a colonoscopy to deliver the filtered donor stool directly into their colon. Additionally, biopsies will be taken during this procedure for routine diagnostic as well as research purposes.

III. Subsequent FMT treatments:

Enemas will be given periodically to complete a total of 1-year therapy.

IV. Follow-up endoscopy and samples:

A similar but more limited procedure (sigmoidoscopy) will be repeated at 14 weeks into the study period. Biopsies will be taken during this procedure for routine diagnostic as well as research purposes.

FMT DONORS:

Potential healthy adult stool donors (between 18 and 45 years of age) will be recruited by the research staff. They will be asked to volunteer for the screening and regularly supply stool samples according to the study protocol.

ELIGIBILITY:
Patient Inclusion Criteria:

* Patients must have a diagnosis of ulcerative colitis based on clinical symptoms, as well as laboratory and colonoscopic findings, including histopathologic results of the intestinal mucosa.
* Pediatric Ulcerative Colitis Activity Index (PUCAI) < 35 [mild activity] as assessed within 4 weeks prior to enrollment and clinical symptoms that are at least stable.
* Patients must be "immunomodulator dependent," i.e., have a history of steroid dependency (lack of clinical remission for over 8 weeks without steroid therapy), and/or being immunomodulator (azathioprine, 6-mercaptopurine, methotrexate, etc.) treated, and/or biologic agent (infliximab, adalimumab, etc.) treated
* Patients ≥ 12 and < 21 years of age are eligible for this trial.
* Patients must be willing to be off current UC therapies.
* Willingness to undergo a surgical consultation prior to FMT treatment.
* Patients who are not enema trained will be required to undergo enema training prior to the start of FMT treatment.
* All patients and/or their parents or legally authorized representatives must sign a written informed consent document. Assent, when appropriate, will be obtained according to institutional guidelines.

Patient Exclusion Criteria:

* Patients who are known to have the following will be excluded:

  1. Decompensated liver cirrhosis (bleeding varices, ascites, encephalopathy or icterus)
  2. Human immunodeficiency virus (HIV)/acquired immune deficiency syndrome (AIDS)
  3. Bone marrow transplantation within the past 150 days
  4. Other severe immunodeficiency
* Patients with severe prior allergic reaction to food will be excluded from the protocol.
* Patients who are pregnant or lactating will be excluded from the protocol.

Donor Inclusion Criteria:

* ≥ 18 years and < 45 years
* Willing to provide stool and blood samples for laboratory testing.
* Body mass index < 30
* Willing to fill out a detailed health screening questionnaire

Ages: 12 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 6 (Actual)
Dates: Start 2014-02; Primary Completion 2014-12 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Assess safety of FMT treatment by recording the frequency of adverse events. | 12 months
  To determine the safety and associated toxicities of serial FMTs in pediatric UC following withdrawal from standard therapy.

SECONDARY OUTCOMES:
Assess efficacy of FMT treatment with the aid of the Pediatric Ulcerative Colitis Activity (PUCAI) Index, a validated measure of clinical disease severity. | 1 year
  To preliminarily assess the efficacy of FMT in inducing or maintaining clinical remission of UC.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Kellermayer, MD, Principal Investigator — Baylor College of Medicine - Texas Children's Hospital
Locations (1):
- Texas Children's Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No